CLINICAL TRIAL: NCT02374658
Title: The Royal Conservatory's ARTS-REHAB Project Research Study
Brief Title: The ARTS-REHAB Project Research Study
Acronym: ARTS-REHAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Royal Conservatory of Music (Other)
Collaborators: Ontario Trillium Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 123123
Record Dates: First submitted 2015-02-23; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Social Wellness Through Engagement in a Creative Process; Patient Engagement
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arts Intervention (Experimental): This group will receive the weekly one-hour Living Through the Arts program in addition to their standard program of rehabilitation activities
  Interventions: Behavioral: Living Through the Arts Intervetion
- Control Group (No Intervention): This group of patients will only receive their standard program of rehabilitation activities

INTERVENTIONS:
Behavioral: Living Through the Arts Intervetion — A weekly one-hour creative arts program that will engage participants in several different creative processes, including visual art, music, dance, drama, and creative writing.
  Other Names: Arts Intervention
  Arms: Arts Intervention

SUMMARY:
The ARTS-REHAB Project Research Study examines how meaningful engagement in a creative process might impact inpatients in rehabilitation centres. Participants in this random control trial study will be recruited from a slow-stream rehabilitation patient population. The study intervention will consist of The Royal Conservatory's Living Through the Arts program. Data will be collected using structured and semi-structured questionnaires along with observational logs and focus groups. This study will explore the effects of the program, comparing the intervention and control group participants' sense of hope and optimism for returning to their daily lives, as well as their sense of engagement in their physical recovery.

DETAILED DESCRIPTION:
The question to be answered through the proposed ARTS-REHAB Project Research Study is: how can meaningful engagement in a creative arts program impact the personal and social wellness of patients in rehabilitation? The ARTS-REHAB Project is a random control trial study that aims to describe and interpret the expectations and experiences of patients' evolving sense of self in recovery as informed by their participation in The Royal Conservatory's Living Through the Arts program. Living Through the Arts is an inter-arts program designed to empower individuals and communities through artistic self-expression and creativity. For those patients receiving this arts intervention in addition to their rehabilitation activities, we expect to see a difference in the following primary measures of their evolving sense of self in recovery compared to patients in a control group. That is, we expect to find an increased sense of hope and optimism; increased sense of future purpose; as well as increased engagement in their rehabilitation. In addition, we will also explore potential attending benefit of functional improvements through a measure of an anticipated decrease in patients' length of hospital stay. Given the complexity of the ARTS-REHAB Project, the study is being conducted in two phases: Phase 1 (now completed) was an 8-week pilot study, conducted at West Park Healthcare Centre and Bridgepoint Active Healthcare between July and October 2014. This pilot evaluated strictly the operational feasibility of implementing an arts program and collecting data with a slow-stream rehabilitation patient population. Phase 2 expands on the learning from the pilot study and involves a two-and-a-half-year Random Control Trial (RTC) study with a total of 8 hospitals (including St. Peter's Hospital in Hamilton, four Toronto hospitals, and 3 other hospitals from across the province). Unlike the pilot study of feasibility, the focus of the two-and-a-half-year study is on the research measures of personal and social wellness described above.

As an extension of a growing literature on arts and healthcare, the proposed research contributes to the knowledge of the transformative potential of creative arts programs / interventions in healthcare settings. Perceptual psychologist Rudolph Arnheim wrote that, "by demonstrating what it can do for the distressed, art reminds us what it is meant to do for everybody" (Arnheim,1986, p. 257). Arnheim's observation aptly captures the spirit of the literature on the contributions of creative arts to the health of individuals with illness and disability (Daykin, Byrne, Soteriou, & Sullivan-Marx, 2006 for review; McNiff, 2009; Malchiodi, ed., 2000; Moon, 2008). However, much of this literature focuses on specific art forms as medical therapy for specific illnesses (e.g., dementia, schizophrenia) and specific demographics (seniors, children). There appears to be a need for studies that examine more broadly how engagement in a creative process serves the whole person and not strictly the disability during recovery / treatment. The ARTS-REHAB Project Research Study takes up this approach by exploring recovery not only in terms of patients' physical needs, but also in terms of their emotional and psychological needs for healing and returning to their daily lives and communities.

Given the "whole person" approach of this study, the degree of a patient's engagement in their recovery must be considered. A diverse literature on patient motivation and compliance has shown that patient engagement can play a role in determining the success of their treatment (O'Gorman, 1975; Meichenbaum & Turk, 1987 for review; McClean & Pound, 2000; Skolasky, et al., 2008). Building on this literature, the proposed study will examine the influence of participation in the arts intervention on patients' motivation and perseverance in their rehabilitation treatment.

A third body of literature relevant to this study explores psycho-social indicators of wellbeing in illness/recovery. Within that broad literature, the concept of optimism emerges as playing an important role in coping with stressful life events. Optimism is characterized by an orientation toward the future where positive explanations are offered even for negative outcomes. Simply put, it is the general expectation that good rather than bad will happen (Sheier & Carver, 1985). According to the literature, optimism has been associated with improved quality of life in the form of lower anxiety/depression for cancer patients (Carver, Pozo, Harris, 1993; Applebaum et al, 2014) and patients with traumatic brain injury (Peleg, et al., 2009), greater satisfaction with a treatment regime for patients suffering myocardial infarction (Barry, et al., 2007), and lower suicidal ideation for university students (Range & Penton, 1994). Much of the optimism literature, however, tends to focus on patients with traumatic chronic illness or mental illness (Eisner, et al., 2009; Johnson, et al., 2009). There is room to build on the evidence with a different patient population, namely, patients undergoing physical rehabilitation. Furthermore, there is room to explore optimism in the context of a specifically arts-based intervention, over and above the prescribed medical treatment.

For the past ten years, the Living Through the Arts program has successfully served different demographic communities (e.g. seniors with dementia, homeless or low income individuals, people with mental illnesses or intellectual disabilities) across Ontario. In keeping with the Living Through the Arts program, the ARTS-REHAB Project will use a variety of art forms and a curriculum of storytelling to help patients in rehabilitation imagine and creatively express their path to recovery in a manner that promotes a strong sense of personal capacity and meaning. More specifically, the curriculum for the ARTS-REHAB Project arts program will consist of themes of health, recovery, and new identities that enable patients to create new stories, shape their sense of purpose, and generate positive images of the future.

The expected outcomes for participants in the arts program of the study include generating: a greater increase in optimism for their recovery; a positive outlook for the future; and a shorter length of stay in hospital when compared to patients who were not involved in the arts program.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants must be health care centre inpatients with an average expected length of stay of 30 days or longer;
2. Eligible participants need to be able to speak, understand, and write English; eligible participants also need to be cognitively able to understand and give written consent and complete research questionnaires (either independently or with minimal assistance);
3. Eligible participants are willing and able to take part in either the intervention group (Living Through the Arts programming) or in the control group;
4. Eligible participants were either community-dwelling or have had a short stay in acute care (no longer than 4 weeks) prior to admission;
5. Eligible participants who are anticipated to return to their homes/communities (or to continue with their rehabilitation as outpatients) following their reconditioning rehabilitation.

Exclusion Criteria:

* early patient discharge (prior to the completion of minimum number of 4 sessions);
* inability of patient to complete questionnaires (due to physical pain or cognitive decline);
* transfer of patient to acute care (without return to slow-stream rehabilitation); and
* (anticipated) transfer of patient to long-term care following rehabilitation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Hope and optimism measured through pre- and post- program questionnaires | 30 - 90 days
  Primary outcome will be measured through pre- and post- program questionnaires administered upon patient intake and prior to patient discharge.
Future purpose measured through pre- and post- program questionnaires | 30 - 90 days
  Primary outcome will be measured through pre- and post- program questionnaires administered upon patient intake and prior to patient discharge
patient engagement measured through pre- and post- program questionnaires | 30-90 days
  Primary outcome will be measured through pre- and post- program questionnaires administered upon patient intake and prior to patient discharge

SECONDARY OUTCOMES:
Length of stay | 30-90 days
  Difference scores will be calculated using patient admission and discharge dates (both anticipated and actual discharge dates).

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Conservatoy of Music, Toronto, Ontario, Canada